CLINICAL TRIAL: NCT06745167
Title: Comparative Efficacy and Safety of Electro-Anatomical Guided Pulsed Field Ablation Versus Radiofrequency Ablation in the Treatment of Persistent Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: Comparative Efficacy and Safety of Extensive Electro-Anatomical Guided Pulsed Field Ablation Versus Radiofrequency Ablation in Persistent Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Albert Einstein College of Medicine and Montefiore Medical Center (Unknown); Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine (Unknown); Shandong University of Traditional Chinese Medicine (Other); Yuhuan Second People's Hospital (Unknown); Changshu Hospital of Traditional Chinese Medicine (Other); The PLA Navy Anqing Hospital (Unknown); Jinan People's Hospital (Unknown); Xuzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, MD, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXT-III
Record Dates: First submitted 2024-11-25; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; pulsed field ablation; radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed field ablation (Experimental): Utilizing pulsed field ablation (PFA), combining pulmonary vein isolation (PVI) with extensive ablation based on anatomical landmarks (including posterior wall box isolation) and electrogram-guided ablation, aiming to target all potential arrhythmic substrates.
  Interventions: Procedure: Pulsed field ablation
- Radiofrequency Ablation (Active Comparator): Using conventional radiofrequency ablation technology, combines pulmonary vein isolation (PVI) with extensive ablation based on anatomical landmarks (including posterior wall box isolation) and electrogram-guided ablation, aiming to target all potential arrhythmic substrates.
  Interventions: Procedure: Radiofrequency ablation alone

INTERVENTIONS:
Procedure: Pulsed field ablation — Utilizing pulsed field ablation (PFA), combining pulmonary vein isolation (PVI) with extensive ablation based on anatomical landmarks (including posterior wall box isolation) and electrogram-guided ablation.
  Arms: Pulsed field ablation
Procedure: Radiofrequency ablation alone — Using conventional radiofrequency ablation technology, combines pulmonary vein isolation (PVI) with extensive ablation based on anatomical landmarks (including posterior wall box isolation) and electrogram-guided ablation
  Arms: Radiofrequency Ablation

SUMMARY:
This multicenter, randomized controlled trial aims to compare the efficacy and safety of extensive electro-anatomical guided pulsed field ablation (EXT-PFA) with traditional radiofrequency ablation (RF) in treating persistent atrial fibrillation (PeAF). The trial seeks to determine if EXT-PFA, which integrates anatomical and electrogram-guided strategies, can provide superior outcomes in terms of safety and effectiveness compared to the standard RF ablation approach.

ELIGIBILITY:
Inclusion Criteria:

1.Adults aged 18-80 years diagnosed with persistent atrial fibrillation. 2.Ineffectiveness or intolerance to at least one Class I or III anti-arrhythmic drug.

Exclusion Criteria:

1. Major valvular diseases needing surgical intervention.
2. Presence of a left atrial thrombus on recent imaging.
3. Recent myocardial infarction or severe heart failure (LVEF ≤ 30%).
4. Current Severe Infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Arrhythmia Recurrence at 12 Months | 12 months after ablation procedure
  Proportion of participants free from atrial fibrillation/atrial flutter/atrial tachycardia recurrence at 12 months post-ablation.

SECONDARY OUTCOMES:
Procedural Safety | From enrollment to completion of follow-up（at least 12 months）
  Incidence of procedural complications such as esophageal injury and pulmonary vein stenosis.
Symptom Relief (EHRA scores) | From enrollment to completion of follow-up（at least 12 months）
  Improvement in clinical symptoms (EHRA scores)
Quality of Life (Short Form 36 Health Survey). | From enrollment to completion of follow-up（at least 12 months）
  quality of life measurements (Short Form 36 Health Survey).
Atrial Fibrillation Burden Reduction | From enrollment to completion of follow-up（at least 12 months）
  Reduction in atrial fibrillation burden assessed through follow-up evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Liu, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- No. 241, West Huaihai Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF